CLINICAL TRIAL: NCT02210832
Title: Financial Incentives for Smoking Cessation Among Disadvantaged Pregnant
Brief Title: Financial Incentives for Smoking Cessation Among Disadvantaged Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stephen T. Higgins, PhD, Professor of Psychiatry and Psychology, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01HD075669-01 (NIH); R01HD075669-01 (NIH)
Record Dates: First submitted 2014-07-31; First posted 2014-08-07 (Estimated); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-05

CONDITIONS: Cigarette Smoking
Keywords: smoking; pregnancy; cessation; incentives
MeSH Terms: conditions — Cigarette Smoking; Smoking | interventions — Practice Guidelines as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Best practices for pregnant smokers (Experimental): Five As plus referral to pregnancy-specific tobacco quit line
  Interventions: Behavioral: Best practices
- Best practices plus financial incentives (Experimental): Best practices plus providing financial incentives contingent on biochemically verified abstinence. Incentives are in the form of vouchers exchangeable for retail items and available through 12-weeks postpartum.
  Interventions: Behavioral: Best practices; Behavioral: financial incentives
- Never-smoker comparison condition (No Intervention): We will follow a group of never-smoker pregnant women matched to smokers on key sociodemographic and obstetrical characteristics for purposes of comparisons in birth/health outcomes at delivery and through 1 year postpartum

INTERVENTIONS:
Behavioral: Best practices
  Other Names: Five As plus referral to pregnancy-specific quit line
  Arms: Best practices for pregnant smokers; Best practices plus financial incentives
Behavioral: financial incentives — financial incentives provided contingent on biochemically confirmed smoking abstinence
  Other Names: contingency management
  Arms: Best practices plus financial incentives

SUMMARY:
Investigators will examine whether adding financial incentives to current best practices for smoking cessation during pregnancy (i.e., referral to pregnancy-specific counseling using a telephone quit line) increases cessation rates and improves infant health. While more expensive upfront compared to best practices alone, the investigators hypothesize that this treatment approach will be economically justified by the later cost savings associated with more women quitting, having healthier babies, and needing less healthcare. It should also help to reduce the greater risk for health problems often seen among those who less well off economically.

DETAILED DESCRIPTION:
Smoking during pregnancy is the leading preventable cause of poor pregnancy outcomes in the U.S. Most pregnant smokers continue smoking through pregnancy producing serious immediate and longer-term adverse health consequences for the infant. Smoking during pregnancy is highly associated with economic disadvantage and a substantive contributor to health disparities.

Efficacious interventions are available, but cessation rates are low (<20%) and improvements in birth outcomes often modest or absent. Current treatments usually entail relatively brief, lower-cost interventions (e.g., pregnancy specific quit lines). There is broad consensus that more effective interventions are sorely needed. This team of investigators has developed a novel behavioral economic intervention in which women earn financial incentives contingent on smoking abstinence. In a metaanalysis of treatments for smoking during pregnancy, effect sizes achieved with financial incentives were several fold larger than those achieved with lower intensity approaches or medications. The intervention also appears to improve birth outcomes and increase breastfeeding duration. While highly promising, further research is needed in at least three areas. (1) The evidence on birth outcomes and breastfeeding is from studies that combined data across trials rather than a single prospective trial, (2) whether the intervention produces other postpartum improvements in health has not been investigated, and (3) the overall cost-effectiveness of this approach has not been examined.

To examine these unanswered questions, the investigators are proposing a randomized, controlled clinical trial comparing the efficacy and cost effectiveness through one year postpartum of current best practices for smoking cessation during pregnancy vs. best practices plus financial incentives among 230 pregnant, Medicaid recipients. A third condition of 115 pregnant nonsmokers matched to the smokers on sociodemographic and health conditions will be included as well to compare the extent to which the treatments reduce the burden of smoking and to estimate how much more might be accomplished by further improvements in this incentives intervention without exceeding cost-effectiveness.

The investigators hypothesize that best practices plus financial incentives will be more effective than usual care practices alone, that the incentives intervention will be cost effective, and that while adding the incentives reduces a greater proportion of the health and economic burden of smoking than best practices alone, more can be done while remaining cost effective.

Overall, the proposed study has the potential to substantially advance knowledge on cost-effective smoking cessation for pregnant women. Importantly, because of the strong association between smoking during pregnancy and economic disadvantage, the proposed study also has the potential to contribute new knowledge relevant to reducing the serious challenges of health disparities.

ELIGIBILITY:
Inclusion Criteria for two intervention arms:

* report being smokers at the time that they learned of the current pregnancy;
* report smoking in the 7 days prior to the first prenatal care visit with biochemical verification;
* < 25 weeks gestation;
* English speaking;
* plan on remaining in the geographical area through 12months postpartum.

Inclusion Criteria for never-smoker comparison condition:

* report being nonsmokers at the time they learned of the current pregnancy;
* report no smoking in the past 6 month;
* Biochemical verification of non-smoker status;
* report smoking < 100 cigarettes in their lifetime;

Exclusion criteria:

* > 25 weeks gestation;
* unavailable for routine assessments through 1 year postpartum;
* opioid substitution therapy;
* untreated/unstable serious mental illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2014-01-31; Primary Completion 2019-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen T Higgins, PhD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, University Health Center Campus, Burlington, Vermont, United States

REFERENCES:
- [Background] Higgins ST, Washio Y, Heil SH, Solomon LJ, Gaalema DE, Higgins TM, Bernstein IM. Financial incentives for smoking cessation among pregnant and newly postpartum women. Prev Med. 2012 Nov;55 Suppl(Suppl):S33-40. doi: 10.1016/j.ypmed.2011.12.016. Epub 2011 Dec 27. PMID 22227223
- [Derived] Shepard DS, Slade EP, Nighbor TD, DeSarno MJ, Roemhildt ML, Williams RK, Higgins ST. Economic analysis of financial incentives for smoking cessation during pregnancy and postpartum. Prev Med. 2022 Dec;165(Pt B):107079. doi: 10.1016/j.ypmed.2022.107079. Epub 2022 May 6. PMID 35533885
- [Derived] Higgins ST, Nighbor TD, Kurti AN, Heil SH, Slade EP, Shepard DS, Solomon LJ, Lynch ME, Johnson HK, Markesich C, Rippberger PL, Skelly JM, DeSarno M, Bunn J, Hammond JB, Roemhildt ML, Williams RK, O'Reilly DM, Bernstein IM. Randomized Controlled Trial Examining the Efficacy of Adding Financial Incentives to Best practices for Smoking Cessation Among pregnant and Newly postpartum Women. Prev Med. 2022 Dec;165(Pt B):107012. doi: 10.1016/j.ypmed.2022.107012. Epub 2022 Mar 3. PMID 35248683

RESULTS

PARTICIPANT FLOW:
Groups:
- Best Practices for Pregnant Smokers: Five As plus referral to pregnancy-specific tobacco quit line
  Best practices
- Best Practices Plus Financial Incentives: Best practices plus providing financial incentives contingent on biochemically verified abstinence. Incentives are in the form of vouchers exchangeable for retail items and available through 12-weeks postpartum.
  Best practices
  financial incentives: financial incentives provided contingent on biochemically confirmed smoking abstinence
Period: Overall Study
Arm/Group | Best Practices for Pregnant Smokers | Best Practices Plus Financial Incentives | Never-smoker Comparison Condition
Started | 91 | 85 | 81
Completed (Defined as completed week-48 postpartum assessment.) | 62 | 49 | 63
Not Completed | 29 | 36 | 18
Not completed — Pregnancy termination . | 3 | 4 | 1
Not completed — Lost to Follow-up | 26 | 32 | 17

BASELINE CHARACTERISTICS:
Population: Women who aborted were removed from the study as per convention in this research area. A total of 8 women were removed for this reason, 3, 4, and 1 in Best practices for pregnant smokers, Best practices plus financial incentives, and Never-smoker comparison conditions.
Groups:
- Total: Total of all reporting groups
Arm/Group | Best Practices for Pregnant Smokers | Best Practices Plus Financial Incentives | Never-smoker Comparison Condition | Total
Number analyzed (Participants) | 88 | 81 | 80 | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (5.5) | 25.4 (5.0) | 25.6 (5.0) | 25.87 (5.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 81 | 80 | 249
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 82 | 74 | 72 | 228
  Unknown or Not Reported | 6 | 7 | 8 | 21
Region of Enrollment [Number; unit: participants]
  United States | 88 | 81 | 80 | 249
Cigarettes smoked per day pre-pregnancy [Mean (Standard Deviation); unit: cigarettes/day] | 18.27 (9.42) | 19.25 (9.87) | 0 (0) | 12.51 (6.43)
Cigarettes smoked per day at 1st antepartum visit [Mean (Standard Deviation); unit: cigarettes/day] | 9.92 (6.18) | 8.99 (5.21) | 0 (0) | 6.30 (3.80)
Age started smoking (yrs) [Mean (Standard Deviation); unit: years] | 15.47 (2.96) | 15.10 (2.92) | 0 (0) | 10.19 (1.96)
% living with other smokers [Count of Participants; unit: Participants] | 68 | 64 | 18 | 150
% with no smoking allowed in home [Count of Participants; unit: Participants] | 62 | 55 | 73 | 190
% with none or few family who smoke [Count of Participants; unit: Participants] | 23 | 20 | 62 | 105
% attempted to quit prepregnancy [Count of Participants; unit: Participants] | 64 | 57 | 0 | 121
# quit attempts during pregnancy [Mean (Standard Deviation); unit: attempts] | 0.73 (2.35) | 0.57 (0.97) | 0 (0) | 0.43 (1.11)
Minnesota Nicotine Withdrawal Scale total score; scale: 0 (none) to 4 (severe);average item scores [Mean (Standard Deviation); unit: scores on a scale] — Minnesota Nicotine Withdrawal Scale We report mean Total Scores (minimum = 0 [no discomfort], maximum = 4 [severe discomfort]) There are 8 scale items, each is scored 0 to 4. Total Scores reflect the average of the eight items.
  We report the average the average Total Score and standard deviation in each treatment condition.
  scores on a scale | 1.60 (0.75) | 1.37 (0.76) | 0 (0) | 0.99 (0.50)
Fagerstrom Test for Nicotine Dependence [Mean (Standard Deviation); unit: 0-10 scale] — The Fagerstrom Test for Nicotine Dependence is a 6-item scale Four items are scored Yes-No with Yes = 1 and No = 0. Two items have four response options each scored 1-4 with lower scores indicating less dependence Items are summed for each test taker to get a total score with a range of 0 (no dependence) to 10 (intense dependence).
  We report the average participant score and standard deviation for each treatment condition.
  0-10 scale | 4.33 (2.30) | 3.98 (2.07) | 0 (0) | 2.77 (1.46)
% endorsing that smoking will greatly harm baby [Count of Participants; unit: Participants] — Item is scored on 0 (not at all) to 4 (a lot); there is a "don't know" item that is recoded as missing. Scale is dichotomized by collapsing items 1-3 vs. 4. We report the number of participants indicating a score of 4.
  Participants | 70 | 69 | 79 | 218
Stress rating scale for past week from 0 (none) to 10 (extreme) [Mean (Standard Deviation); unit: Scores on a scale] — This is a single item scale on which each participant rates their past week's stress as 0 (none) to 10 (extreme). We report the mean score and standard deviation for each treatment condition.
  Scores on a scale | 6.3 (2.2) | 5.0 (2.5) | 3.3 (2.1) | 4.9 (2.3)
Beck Depression Inventory total score [Mean (Standard Deviation); unit: units on a 0-63 scale] — The Beck Depression Inventory contains items 21 items each scored 0 (least) to 3 (most). Item scores are summed for a total score ranging from 0-63. We report the mean total score and standard deviation for each treatment condition.
  units on a 0-63 scale | 12.8 (8.6) | 10.0 (7.4) | 5.8 (5.2) | 9.5 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence Abstinence Levels at Final Antepartum Assessment
Description: Abstinence was defined as woman reports that she has not smoked, not even a puff, in the past 7 days and self-report is biochemically verified via urine cotinine testing
Time Frame: collected once per women at approximately 28-weeks gestation in each of the two smoking arms
Population: Comparison of women in two smoking-cessation arms
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practices for Pregnant Smokers | Best Practices Plus Financial Incentives
Number analyzed (Participants) | 88 | 81
Participants | 8 | 31
Statistical Analysis 1: Comparison: Best Practices for Pregnant Smokers vs Best Practices Plus Financial Incentives; Hypothesized that women assigned to Best practices plus financial incentives would achieve greater abstinence than women assigned to Best practices only; Test type: Superiority — 38.27% vs. 9.09%; p < 0.001, Chi-squared — p value is not adjusted for multiple comparisons. A priori threshold for significance was P < 0.05; chi square test statistic = 20.23, df = 1

2. Secondary Outcome: 7-day Point Prevalence Abstinence Postpartum
Description: Compare two treatment arms on 7-day point-prevalence abstinence assessed at 2-, 4-, 8-, 12-, 24- and 48-weeks postpartum. Abstinence was defined as self-report of no smoking in past 7 days, not even a puff, with biochemical verification of self-report using urine cotinine testing
Time Frame: Repeated assessments completed at 2-, 4-, 8-, 12-, 24-, and 48-weeks postpartum
Population: Hypothesized that women assigned to Best practices plus financial incentives would achieve greater smoking abstinence than women assigned to Best practices only.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practices for Pregnant Smokers | Best Practices Plus Financial Incentives
Number analyzed (Participants) | 88 | 81
Participants
  2 weeks postpartum | 17 | 31
  4 weeks postpartum | 14 | 30
  8 weeks postpartum | 12 | 25
  12 weeks postpartum | 10 | 21
  24 weeks postpartum | 11 | 14
  48 weeks postpartum | 10 | 13
Statistical Analysis 1: Comparison: Best Practices for Pregnant Smokers vs Best Practices Plus Financial Incentives; Test type: Superiority; p < 0.05, Chi-squared; Used generalized estimating equation utilizing a logistic link function with treatment condition and assessment time adjusting for covariates
Statistical Analysis 2: Comparison: Best Practices for Pregnant Smokers vs Best Practices Plus Financial Incentives; Trial condition by assessment time interaction; Test type: Superiority; p = 0.003, Mixed Models Analysis — chi square test statistic = 21.93, df=7; Conducted a generalized estimating equation utilizing a logistic link function with treatment condition and assessment time adjusting for covariates

3. Secondary Outcome: Breastfeeding in the Three Trial Arms
Description: Compare the three trial arms on overall percentage of women continuing to breastfeed at repeated postpartum assessments
Time Frame: Repeated assessments completed at 2-, 4-, 8-, 12-, 24-, and 48-weeks postpartum
Population: Breastfeeding data were not obtained on all women. The number of women with at least one assessment with breastfeeding data in each group is: Best practices = 79, Best practices plus financial incentives = 69, Never-Smokers = 78
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practices for Pregnant Smokers | Best Practices Plus Financial Incentives | Never-smoker Comparison Condition
Number analyzed (Participants) | 79 | 69 | 78
Participants
  2-weeks postpartum | 49 | 50 | 59
  4-weeks postpartum | 40 | 40 | 56
  8-weeks postpartum | 34 | 34 | 48
  12-weeks postpartum | 28 | 28 | 43
  24-weeks postpartum | 21 | 21 | 36
  48-weeks postpartum | 9 | 9 | 23
Statistical Analysis 1: Comparison: Best Practices for Pregnant Smokers vs Best Practices Plus Financial Incentives vs Never-smoker Comparison Condition; Interaction of trial condition and time; Test type: Superiority; p = 0.48, Mixed Models Analysis — chi square test statistic = 9.52, df = 10; [statistical method as in outcome 2, analysis 2]

4. Secondary Outcome: Breastfeeding While Abstinent From Smoking
Description: We compared the three trial arms on the percent of women who reported breastfeeding and were biochemically confirmed to be abstinent from smoking at each postpartum assessment.
Time Frame: Repeated assessments completed at 2-, 4-, 8-, 12-, 24-, and 48-weeks postpartum
Population: Comparing women in each trial condition who reported breastfeeding and were biochemically confirmed abstinent from smoking at each postpartum assessment. Breastfeeding data were not obtained on all women. The number of women with at least one assessment with breastfeeding data in each group is: Best practices = 79, Best practices plus financial incentives = 69, Never-Smokers = 78
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practices for Pregnant Smokers | Best Practices Plus Financial Incentives | Never-smoker Comparison Condition
Number analyzed (Participants) | 79 | 69 | 78
Participants
  2-weeks postpartum | 15 | 29 | 59
  4-weeks postpartum | 11 | 24 | 56
  8-weeks postpartum | 9 | 19 | 48
  12-weeks postpartum | 7 | 15 | 43
  24-weeks postpartum | 7 | 9 | 36
  48-weeks postpartum | 3 | 5 | 23
Statistical Analysis 1: Comparison: Best Practices for Pregnant Smokers vs Best Practices Plus Financial Incentives vs Never-smoker Comparison Condition; Examining main effect of treatment condition; Test type: Superiority; p < 0.0001, Mixed Models Analysis — chi square test statistic = 33.51, df = 2; [statistical method as in outcome 2, analysis 2]
Statistical Analysis 2: Comparison: Best Practices for Pregnant Smokers vs Best Practices Plus Financial Incentives vs Never-smoker Comparison Condition; Testing interaction of treatment condition and assessment time; Test type: Superiority; p = 0.89, Mixed Models Analysis — chi square test statistic = 5.00, df = 10

5. Secondary Outcome: Craving Item From the Minnesota Nicotine Withdrawal Scale (MNWS).
Description: The craving item is on a 0 (none) to 4 (severe) scale. We report mean (SEM) scores.
Time Frame: Outcomes reported for 8 assessments (early pregnancy, late pregnancy, 2, 4, 8, 12, 24, 28 weeks postpartum.
Population: Comparing between women assigned to the two smoking-cessation trial conditions.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Best Practices for Pregnant Smokers | Best Practices Plus Financial Incentives
Number analyzed (Participants) | 88 | 81
scores on a scale
  early antepartum | 2.73 (0.14) | 1.75 (0.15)
  late antepartum | 2.30 (0.14) | 1.52 (0.15)
  2 weeks postpartum | 2.14 (0.15) | 1.39 (0.16)
  4 weeks postpartum | 2.17 (0.15) | 1.55 (0.16)
  8 weeks postpartum | 2.27 (0.15) | 1.75 (0.16)
  12 weeks postpartum | 2.33 (0.14) | 1.72 (0.16)
  24 weeks postpartum | 1.97 (0.15) | 1.97 (0.16)
  48 weeks postpartum | 2.10 (0.16) | 1.99 (0.17)
Statistical Analysis 1: Comparison: Best Practices for Pregnant Smokers vs Best Practices Plus Financial Incentives; Test type: Superiority; p < 0.001, Mixed Models Analysis; Method was mixed model repeated measures analysis of covariance

6. Secondary Outcome: Nicotine Withdrawal Total Scores for the Two Smoking-cessation Trial Conditions.
Description: Reporting mean total scores and SEM from the Minnesota Nicotine Withdrawal Scale (MNWS). Total score is an average of 7 items, with each item on a 0 (none) to 4 (severe) scale.
Time Frame: Outcomes reported for 8 assessments (early pregnancy, late pregnancy, 2, 4, 8, 12, 24, 28 weeks postpartum.
Population: Comparing women assigned to the two smoking-cessation trial conditions.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Best Practices for Pregnant Smokers | Best Practices Plus Financial Incentives
Number analyzed (Participants) | 88 | 81
scores on a scale
  Early antepartum | 1.47 (0.08) | 1.02 (0.08)
  Late antepartum | 1.38 (0.08) | 0.93 (0.08)
  2-weeks postpartum | 0.80 (0.08) | 0.70 (0.09)
  4-weeks postpartum | 0.80 (0.08) | 0.68 (0.09)
  8-weeks postpartum | 0.92 (0.08) | 0.68 (0.08)
  12-weeks postpartum | 0.86 (0.08) | 0.59 (0.08)
  24-weeks postpartum | 0.81 (0.08) | 0.78 (0.09)
  48-weeks postpartum | 1.03 (0.8) | 0.84 (0.09)
Statistical Analysis 1: Comparison: Best Practices for Pregnant Smokers vs Best Practices Plus Financial Incentives; Examine interaction of treatment condition and assessment time; Test type: Superiority; p < 0.001, ANCOVA — F[7,922]=3.62; Repeated measures analysis of covariance was conducted with Bonferroni corrections for post-doc tests and across repeated assessments
Statistical Analysis 2: Comparison: Best Practices for Pregnant Smokers vs Best Practices Plus Financial Incentives; Test type: Superiority; p < 0.001, Mixed Models Analysis; Method was mixed model repeated measures analysis of covariance

7. Secondary Outcome: Infant Growth in First Year of Life
Description: Infant growth (length & weight) expressed a Body Mass Index (BMI) percentile score was assessed at delivery, 24- and 48-week postpartum assessments.
Time Frame: delivery, 24-week, and 50-week postpartum assessments
Population: There was data available for one or more assessments for 79, 67, and 77 of infants born to mothers in the Best practices, Best practices plus financial incentives, and never-smoker conditions. We compared body mass index (BMI) percentile scores between infants from the three trial conditions at delivery, 24-weeks postpartum, and 48-weeks postpartum.
Measure: Mean (Standard Error); unit: BMI Percentile
Arm/Group | Best Practices for Pregnant Smokers | Best Practices Plus Financial Incentives | Never-smoker Comparison Condition
Number analyzed (Participants) | 79 | 67 | 77
BMI Percentile
  Birth | 31.39 (3.35) | 34.92 (3.51) | 40.56 (3.20)
  24-weeks postpartum | 56.19 (3.36) | 59.14 (3.71) | 46.15 (3.39)
  48-weeks postpartum | 65.97 (3.73) | 65.69 (4.06) | 66.62 (3.47)
Statistical Analysis 1: Comparison: Best Practices for Pregnant Smokers vs Best Practices Plus Financial Incentives vs Never-smoker Comparison Condition; Test type: Superiority; p = 0.009, Mixed Models Analysis; Method was mixed model repeated measures analysis of covariance

8. Secondary Outcome: Birth Outcomes (% Small for Gestational Age Deliveries)
Description: Birth outcomes were compared between the three study arms. Small for gestational age was defined as <10th percentile using INTERGROWTH-21st [2021] https://intergrowth21.tghn.org/about/about-us/.
Time Frame: delivery
Population: Comparison of three trial conditions on SGA deliveries
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practices for Pregnant Smokers | Best Practices Plus Financial Incentives | Never-smoker Comparison Condition
Number analyzed (Participants) | 88 | 76 | 79
Participants
  Small for Gestational Age | 16 | 8 | 2
  Normal size for gestational age | 72 | 68 | 77
Statistical Analysis 1: Comparison: Best Practices for Pregnant Smokers vs Best Practices Plus Financial Incentives vs Never-smoker Comparison Condition; Test type: Superiority; p = 0.01, Regression, Logistic; Method is logistic regression adjusted for covariates

9. Secondary Outcome: Birth Outcomes (Percent Preterm [<37 Weeks] Deliveries)
Description: Compared the three trials conditions on preterm deliveries.
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practices for Pregnant Smokers | Best Practices Plus Financial Incentives | Never-smoker Comparison Condition
Number analyzed (Participants) | 88 | 76 | 79
Participants
  preterm | 6 | 10 | 6
  >/= 37 weeks | 82 | 66 | 73
Statistical Analysis 1: Comparison: Best Practices for Pregnant Smokers vs Best Practices Plus Financial Incentives vs Never-smoker Comparison Condition; Test type: Superiority; p < 0.05, Chi-squared

10. Secondary Outcome: Birth Outcomes (NICU Admissions)
Description: Compared three trial conditions on percent of NICU admissions
Time Frame: at delivery
Population: Compared three trial conditions on NICU admissions.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practices for Pregnant Smokers | Best Practices Plus Financial Incentives | Never-smoker Comparison Condition
Number analyzed (Participants) | 88 | 76 | 79
Participants
  NICU admitted | 11 | 10 | 11
  no NICU | 77 | 66 | 68
Statistical Analysis 1: Comparison: Best Practices for Pregnant Smokers vs Best Practices Plus Financial Incentives vs Never-smoker Comparison Condition; Test type: Superiority; p < 0.05, Chi-squared

11. Secondary Outcome: Ages & Stages Questionnaire (ASQ)
Description: The ASQ assesses infant development in five areas (communication [Comm], gross motor [GM], fine motor [FM], problem solving [PrbSlv], personal-social [PerSoc]); Each area includes six items, each with a possible value of 0, 5, 10, along with a cutoff to dichotomize infants into typical/normal vs. monitor/potential delay categories for an area. Scores in each area are compared to norms; scores with 1 standard deviation of the norm mean are categorized as typical/normal and those greater than one standard deviation below the norm mean are categorized as monitor/potential delay. We report the dichotomized outcomes for each of the six areas at the 24-week and 48-week assessments noting the number of infants in each treatment condition in the monitor/potential delay category.
Time Frame: 24- and 48-weeks postpartum
Population: Overall number of participants analyzed represents the number of participants for whom we obtained data on this outcome at 24-weeks postpartum; at 48-weeks the overall number analyzed were 69, 56, and 72 in Best Practices, Best Practices plus financial incentives, and never-smokers, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practices for Pregnant Smokers | Best Practices Plus Financial Incentives | Never-smoker Comparison Condition
Number analyzed (Participants) | 72 | 58 | 68
Participants
  Comm at 24-weeks | 1 | 2 | 3
  Comm at 48-weeks | 2 | 0 | 3
  GM at 24-weeks | 18 | 10 | 10
  GM at 48-weeks | 14 | 6 | 13
  FM at 24-weeks | 28 | 17 | 16
  FM at 48-weeks | 7 | 5 | 7
  PrbSlv at 24-weeks | 17 | 7 | 10
  PrbSlv at 48-weeks | 10 | 3 | 13
  PerSoc at 24-weeks | 15 | 9 | 13
  PerSoc at 48-weeks | 11 | 8 | 9

12. Secondary Outcome: Birth Outcome: Gestational Age at Delivery
Description: Birth outcomes were obtained from the birth record. Gestational age was expressed in weeks.
Time Frame: at delivery
Population: Birth outcomes were obtained from 88, 76, and 79 infants born to women in the best practices, best practices plus financial incentives, and never-smoker conditions.
Measure: Mean (Standard Error); unit: gestational age (weeks)
Arm/Group | Best Practices for Pregnant Smokers | Best Practices Plus Financial Incentives | Never-smoker Comparison Condition
Number analyzed (Participants) | 88 | 76 | 79
gestational age (weeks) | 39.18 (0.22) | 38.69 (0.23) | 39.35 (0.22)
Statistical Analysis 1: Comparison: Best Practices for Pregnant Smokers vs Best Practices Plus Financial Incentives vs Never-smoker Comparison Condition; Test type: Superiority; p < 0.05, ANCOVA

13. Secondary Outcome: Cost Per Participant
Description: Cost per participant for BP+FI and BP interventions. These costs per participant are used in calculation of the Incremental Cost Effectiveness Ratio (ICER). This ICER measure is the added healthcare sector cost per participant for BP+FI compared to BP relative to estimated net health gain per participant (QALY). Maternal net health gains in QALYs from cessation difference between treatment conditions at 24 weeks postpartum were based on Stapleton & West, 2012, Nicotine Tob Res; 14: 463-71.
Time Frame: Trial entry through 24-weeks postpartum (approximately one year following smoking-cessation quit date).
Population: All participants treated in best practices plus financial incentives and best practices trial conditions.
Measure: Mean (Standard Error); unit: U.S. dollars
Groups:
- Best Practices: Best Practices: 5As plus referral to tobacco quit line
Arm/Group | Best Practices Plus Financial Incentives | Best Practices
Number analyzed (Participants) | 81 | 88
U.S. dollars | 23007.01 (1284.83) | 22372.25 (1594.23)

14. Secondary Outcome: Quality of Life Years Gained (QALYs)
Description: Smoking abstinence at the 24-week assessment was converted into quality of life years gained using standardized tables reported in Stapleton & West, 2012, Nicotine Tob Res; 14: 463-71.
Time Frame: 24 weeks postpartum
Population: Analysis of results for this measure cannot be reported separately for each treatment arm. Thus, treatment conditions were combined because the outcome is the difference in quality of life years gained (QALYs) between conditions.
Measure: Mean (Standard Deviation); unit: net years gained
Groups:
- Combined Best Practices and Best Practices Plus Financial Incentives: Best practices: Five As plus referral to pregnancy-specific tobacco quit line
  Best practices plus providing financial incentives contingent on biochemically verified abstinence. Incentives are in the form of vouchers exchangeable for retail items and available through 12-weeks postpartum.
Arm/Group | Combined Best Practices and Best Practices Plus Financial Incentives
Number analyzed (Participants) | 169
net years gained | 0.0267 (0.0412)

15. Secondary Outcome: Incremental Cost Effectiveness Ratio (ICER)
Description: A summary measure representing the economic value of an intervention (BP+FI) compared with an alternative (BP). The measure type used below is 'number' due to the fact that this measure is simply a ratio of mean dollars divided by mean years gained between the treatment conditions. Thus there was no alternative measure type that could be used or measure of dispersion available.
Time Frame: 24 weeks postpartum
Population: Treatment conditions were combined because the ICER outcome is a measure of the economic benefit of the BP+FI intervention relative to the BP comparator.
Measure: Number; unit: dollars per years gained
Arm/Group | Combined Best Practices and Best Practices Plus Financial Incentives
Number analyzed (Participants) | 169
dollars per years gained | 23511

16. Other Pre Specified Outcome: Additional Birth Outcome: Mean Birth Weight
Description: Birth weight was obtained for each infant from the birth record and expressed in grams. We report the group mean and standard error for each treatment condition.
Time Frame: at delivery
Population: Birth outcomes were obtained for 88, 76, and 79 infants of mothers in best practices, best practices plus financial incentives, and never-smokers.
Measure: Mean (Standard Error); unit: weight (grams)
Arm/Group | Best Practices for Pregnant Smokers | Best Practices Plus Financial Incentives | Never-smoker Comparison Condition
Number analyzed (Participants) | 88 | 76 | 79
weight (grams) | 3176.39 (46.74) | 3214.84 (50.11) | 3391.14 (49.64)
Statistical Analysis 1: Comparison: Best Practices for Pregnant Smokers vs Best Practices Plus Financial Incentives vs Never-smoker Comparison Condition; Test type: Superiority; p = 0.006, ANCOVA; All comparisons adjusted for infant gestational age at time of delivery

ADVERSE EVENTS:
Time Frame: On average women were followed for 1 year, 6 months (end of 1st trimester of pregnancy through 1 year postpartum).
Description: We report the number of instances of pregnancy termination/fetal demise per treatment condition.
Arm/Group | Best Practices for Pregnant Smokers | Best Practices Plus Financial Incentives | Never-smoker Comparison Condition
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/85 | 0/81
Serious Adverse Events (participants affected / at risk) | 3/91 | 4/85 | 1/81
Other Adverse Events (participants affected / at risk) | 0/91 | 0/85 | 0/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Best Practices for Pregnant Smokers (N=91) | Best Practices Plus Financial Incentives (N=85) | Never-smoker Comparison Condition (N=81)
Pregnancy termination/fetal demise (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT02210832/Prot_SAP_000.pdf